CLINICAL TRIAL: NCT02807610
Title: Comparison of Induction Characteristics of Two Anaesthetic Agents-Etomidate Lipuro and Propofol
Brief Title: Etomidate vs Propofol-Induction Characteristics
Acronym: Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maharashtra University of Health Sciences (Other)
Responsible Party: Principal Investigator, Shakuntala Basantwani, Associate Professor, Maharashtra University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PS/IEC-HR/DISS/38
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Hemodynamics; Side Effects
Keywords: Etomidate lipuro; Induction characteristics
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV Propofol and IV Etomidate lipuro (Experimental): After premedication with IV midazolam 0.2mg kg-1, IV Fentanyl 2ug kg-1, Group P Patients received IV Propofol 2mg kg-1 slowly over 60 seconds till Entropy of 40 as a comparator agent in patients undergoing Medical termination of pregnancy(MTP) and Group ' E' Patients received IV Etomidate Lipuro 0.3mg kg-1 slowly over 60 seconds till Entropy of 40 as intervention agent in patients undergoing MTP
  Interventions: Drug: Inj Etomidate; Drug: Injection Propofol
- IV Etomidate Lipuro and Placebo (Active Comparator): After premedication with IV midazolam 0.2mg kg-1, IV Fentanyl 2ug kg-1, Group ' E' Patients received IV Etomidate Lipuro 0.3mg kg-1 slowly over 60 seconds till Entropy of 40 as intervention agent in patients undergoing MTP and placebo group received normal saline
  Interventions: Drug: Inj Etomidate; Drug: Placebo for Propofol

INTERVENTIONS:
Drug: Inj Etomidate — Induction of anesthesia using IV Etomidate 0.3mg kg-1 as a single dose in patients undergoing day care procedure, after premedication with IV midazolam 0'.2mg kg-1 and IV Fentanyl 2ug kg-1.
  Other Names: Etomidate Lipuro
Drug: Injection Propofol — Induction of anesthesia using IV Propofol 2mg kg-1 as a single dose in patients undergoing day care procedure, after premedication with IV midazolam 0.2mg kg-1 and IV Fentanyl 2ug kg-1
  Arms: IV Propofol and IV Etomidate lipuro
Drug: Placebo for Propofol — After premedication with IV midazolam 0.2mg/kg and IV Fentanyl 2ug/kg Placebo was given.
  Arms: IV Etomidate Lipuro and Placebo

SUMMARY:
The ideal induction agent for day care surgery should have properties of rapid, smooth induction, better haemodynamic profile, faster recovery and devoid of side effects in the form of pain on injection, involuntary movements, respiratory depression and post-operative nausea/vomiting. Propofol is the drug being used for day care surgeries because of its rapid, smooth induction and faster recovery. But its use is associated with pain on injection (even with added lidocaine), hypotension and respiratory depression. So the need for an agent with better hemodynamic control and lesser side effects was felt. The introduction of etomidate lipuro revolutionised the anaesthesia practice. It possesses many of the properties of an ideal induction agent. This newer formulation of etomidate in lipid emulsion i.e. etomidate lipuro is known to have rapid, smooth induction, haemodynamic stability and lesser side effects than older etomidate with propylene glycol (hypnomidate).

Hence, investigators devised a prospective randomized controlled open trial and compared this newer lipid formulation of etomidate with propofol in terms of - induction time, haemodynamic parameters and side effect profile.

DETAILED DESCRIPTION:
The administration of a suitable drug by intravenous route for induction of anaesthesia has been an important component of anaesthetic management.The ability to deliver safe and effective anaesthesia with minimal side effects and rapid recovery is critically important to ensure safe and early discharge. An ideal intravenous (IV) anaesthetic agent should, have rapid onset, rapid recovery, be without undesirable cardiac and respiratory depression and lesser untoward effects like pain on injection, nausea, vomiting etc.No single drug is ideal.

Propofol (propofol 1%) has a smooth and rapid induction, rapid recovery, cerebro-protective effect but it causes hypotension, bradycardia, respiratory depression pain on injection.Etomidate is a hypnotic agent causing minimal histamine release and very stable hemodynamic profile. In the present study, investigators evaluated the induction characteristics and side effect profile of this newer lipid formulation of etomidate and compared it with propofol in same lipid formulation.

Material and Methods: Hundred ASA I & II patients in the age group 18-60 yrs, scheduled for dilatation and curettage procedure were randomly allocated in two groups based on induction agent Etomidate lipuro or Propofol.

Both groups received intravenous midazolam 0.02mg /kg and fentanyl 2 µg /kg as premedication. After induction with the desired agent titrated to bispectral index Entropy 40, the time to achieve BIS values to 40 (BIS 40 time) were measured. Heart rate, mean arterial pressures were recorded at baseline, induction and upto 10 minutes. Patients were asked for pain at the injection site, postoperative nausea and observed visually for myoclonus, apnea and thrombophlebitis.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II Female patients
* Elective Medical Termination of Pregnancy (MTP) surgery

Exclusion Criteria:

* Hemo-dynamically unstable patients
* Allergic to egg protein
* Patients with epilepsy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Heart rate per minute | Change in Heart rate per minute from baseline value every five minutes for 30 minutes.
  Mean of Heart rate per minute at above mentioned time intervals was measured and any study drug causing bradycardia (Heart rate <50 was noted .
Mean Arterial Pressure | Change in Mean Arterial Pressure(MAP) in mm of Hg from baseline value every 5 minutes for 30 minutes
  Mean value of Mean Arterial Pressures(Summation of MAP divided by number of patients) at above mentioned time intervals was noted and study drug causing Hypotension(MAP< 90mm of Hg) was noted.

SECONDARY OUTCOMES:
Side effects of the drugs in the form of Pain on injection | 2 minutes after injection of study drug.
  0. No pain. I. Verbal complaint of pain. II. Withdrawal of arm. III. Both verbal complaint and withdrawal of arm. 0. No pain. I. Verbal complaint of pain. II. Withdrawal of arm. III. Both verbal complaint and withdrawal of arm. 0. No pain. I. Verbal complaint of pain. II. Withdrawal of arm. III. Both verbal complaint and withdrawal of arm. Pain on injection was measured using scale as 0 no pain,1verbal complaint to pain,2 withdrawal of arm,3 both verbal complaint and withdrawal of arm
Myoclonic movements | 60 seconds after injection of study drug
  Using Myoclonus scale as 0.No myoclonic movement. I. Minor myoclonic movement. II. Moderate myoclonic movement. III. Major myoclonic
Thrombophlebitis | 24 hours postoperatively
  Presence or absence of inflammation of vein through which the drug was injected.

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available.